CLINICAL TRIAL: NCT02108353
Title: Multicenter, Randomized, Double-blind, Placebo Controlled Trial of 2 mg Melatonin for Circadian Phase Adjustment and Improvement of Metabolic Control in Night Shift Workers
Brief Title: Circadian Phase Adjustment and Improvement of Metabolic Control in Night Shift Workers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EuRhythDia II
Record Dates: First submitted 2013-11-04; First posted 2014-04-09 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Sleep Disorders, Circadian Rhythm
Keywords: Type 2 Diabetes; metabolic control; Metabolomics; Circadian Rhythm; Melatonin; Biomarker; Clock Gene; PBMC; Cardiovascular function; Epigenetic modification; Lifestyle Intervention
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Diabetes Mellitus, Type 2 | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin 2mg (Active Comparator): The study medication will be compared to placebo control.
  Interventions: Drug: Melatonin 2mg
- Placebo (Placebo Comparator): The study medication will be compared to placebo control.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin 2mg — once daily, 0.5-1 hours before going to bed and 1-2 hours after the last meal for 12 weeks.
  Other Names: Circadin®
  Arms: Melatonin 2mg
Drug: Placebo — once daily, 0.5-1 hours before going to bed and 1-2 hours after the last meal for 12 weeks.
  Other Names: None active substances
  Arms: Placebo

SUMMARY:
EuRhythDia II is a multicenter, randomized, double-blind controlled study. The rationale of EuRhythdia is to explore the effects of 12 weeks of timed melatonin treatment on circadian rhythm, metabolic control and cardiovascular function in night shift workers. The 12 weeks of intervention will be followed by 12 weeks of washing out.

DETAILED DESCRIPTION:
Modern lifestyle has dramatically changed the daily rhythms of life. Physical activity, diet and light exposure are no longer restricted to daytime hours due to increased shift work. Recent scientific reports have shown that shift work leads to disruption of circadian rhythms and promotes diabetes, obesity and cardiovascular disease. Until now only few studies investigating circadian rhythm disturbances in the context of type 2 diabetes and obesity have been conducted in man. Thus, knowledge of the molecular pathways and the responsibles genes in man are missing and have been identified only in animal studies.

The objective of the project is to achieve breakthroughs in the understanding of the causality between inner clock rhythm disturbances and the development of type 2 diabetes and obesity. The provided data on the interaction between genes, epigenetics, metabolism, cardiovascular function and the internal clock are intended to contribute to identify novel biomarkers and novel therapeutic approaches focusing on circadian rhythms to reduce the occurence of diabetes and obesity in shift worker.

ELIGIBILITY:
Inclusion Criteria:

* Male and female above the age of 18
* Night shift workers on regular night shifts (at least 6 months before inclusion into the study and at least 4 night shifts per month during the study period

Exclusion Criteria:

* pregnancy or breast feeding
* Known autoimmune disease
* Current or relevant history of physical or psychiatric illness
* Evidence of renal insufficiency or liver disease
* Known or suspected intolerance or hypersensitivity to the study medication
* Use of certain drugs within 4 weeks prior to the inclusion to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01; Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Efficacy (AUC) | baseline and 12 weeks
  The change in the area under the curve (AUC) of blood glucose during an oral glucose tolerance test between baseline and 12 weeks of intervention.

SECONDARY OUTCOMES:
Efficacy BMI | baseline, 12 weeks and 24 weeks
  The change in body weight, BMI, abdominal circumference, biomarkers and vascular function between baseline and 12 weeks of intervention and between week 12 and 24.
Efficacy expression pattern of clock genes | baseline, 12 weeks and 24 weeks
  The change in the gene expression patterns of Clock genes in peripheral blood monocytic cells (PBMC) between baseline and 12 weeks of intervention and between week 12 and 24.
Efficacy glucose homeostasis (HOMA-index) | baseline, 12 weeks and 24 weeks
  The change in the HOMA-index (Homeostasis Model Assessment) between baseline and 12 weeks of intervention and between week 12 and 24.
Efficacy glucose homeostasis (QUICKI-index) | baseline, 12 weeks and 24 weeks
  The change in the QUICKI-index (quantitative insulin sensitivity check index) between baseline and 12 weeks of intervention and between week 12 and 24.
Efficacy glucose homeostasis (Stumvoll ISI-index) | baseline, 12 weeks and 24 weeks
  The change in HbA1c between baseline and 12 weeks of intervention and between week 12 and 24.
Efficacy glucose homeostasis (HbA1c) | baseline, 12 weeks and 24 weeks
  The change in the Stumvoll ISI (Stumvoll insulin sensitivity index) between baseline and 12 weeks of intervention and between week 12 and 24.
Efficacy epigenetic profiles | 12 weeks and 24 weeks
  The differences in epigenetic profiles of genes involved in circadian rhythm between the study groups after 12 weeks of intervention and between week 12 and 24.
Efficacy biomarkers | baseline, 12 weeks and 24 weeks
  The differences in plasma and serum biomarkers between baseline and 12 weeks of intervention and between week 12 and 24.
Efficacy AUC Insulin 24 weeks | 12 weeks and 24 weeks
  The change in the area under the curve (AUC) of blood insulin during an oral glucose tolerance test between week 12 and week 24 (= after 12 weeks without intervention).
Efficacy AUC glucose 24 weeks | 12 weeks and 24 weeks
  The change in the area under the curve (AUC) of blood glucose during an oral glucose tolerance test between week 12 and week 24 (= after 12 weeks without intervention).
Efficacy AUC insulin 12 weeks | baseline and 12 weeks
  The change in the area under the curve (AUC) of blood insulin during an oral glucose tolerance test between baseline and 12 weeks of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer H Boeger, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (3):
- Germany (2):
  - University Medical Center Aachen, Aachen, North Rhine-Westphalia
  - CTC North GmbH & Co. KG, Hamburg
- Department of Systems Medicine, Rome, Lazio, Italy

REFERENCES:
- See also: Trial homepage — http://eurhythdia.eu